CLINICAL TRIAL: NCT05690490
Title: Treament for Colorectal Neoplasms by Metod Endoscopic Mucosal Resection With Circumferential Mucosal Incision
Brief Title: Endoscopic Mucosal Resection With Circumferential Incision for Colorectal Neoplasms
Acronym: C-EMR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: State Scientific Centre of Coloproctology, Russian Federation (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 26/20
Record Dates: First submitted 2021-01-18; First posted 2023-01-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Endoscopic Mucosal Resection With Circumferential Incision
Keywords: C-EMR; Endoscopic treatment; colorectal neoplasm; circumferential incision
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Intervention Model Description: prospective, single-center, randomized, non inferiority
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- endoscopic mucosal resection with circumferential incision (Experimental): The endoscope will be passed into the intestine to the site of the tumor. Then, using an endoscopic needle, a solution will be injected into the submucosa to remove the neoplasm. Using an endoscopic knife (insulated tip knife, Olympus or Water Jet, Erbe), a circular incision will be made around the lesion. Then there will be a one-stage electro excision of the neoplasm using an endoscopic loop.
  Interventions: Procedure: Endoscopic mucosal resection with circumferential incision
- endoscopic submucosal dissection (Active Comparator): The endoscope will be passed into the intestine to the site of the tumor. Then, using an endoscopic needle, a solution will be injected into the submucosa to remove the neoplasm. Using an endoscopic knife (Insulated Tip Knife, Olympus or Water Jet, Erbe), the lesion will be resected through the submucosal plane using the eb-block principle, after which the patient will be monitored.
  Interventions: Procedure: Endoscopic submucosal dissection

INTERVENTIONS:
Procedure: Endoscopic mucosal resection with circumferential incision — The endoscope will be passed into the intestine to the site of the tumor. Using an endoscopic needle, the solution will be injected into the submucosa to create a pillow. Then, using an endoscopic knife (insulated tip knife, Olympus or Water Jet, Erbe), a circular incision will be made around the lesion with an offset of 2-5 mm. Then there will be a one-stage electro excision of the neoplasm using an endoscopic loop.
  Arms: endoscopic mucosal resection with circumferential incision
Procedure: Endoscopic submucosal dissection — The endoscope will be passed into the intestine to the site of the tumor. Using an endoscopic needle, the solution will be injected into the submucosa to create a pillow. Then, using an endoscopic knife (insulated tip knife, Olympus or Water Jet, Erbe), a circular incision is made around the lesion. Then dissection will be performed in the submucosal layer.
  Arms: endoscopic submucosal dissection

SUMMARY:
This is a prospective randomized trial to improve the results of treatment of patients with colorectal neoplasms.

DETAILED DESCRIPTION:
Generally, endoscopic mucosal resection (EMR) and endoscopic submucosal dissection (ESD) are the methods of choice for the removal of benign and early malignant neoplasms of the colon. However, there are certain difficulties in terms of the EMR technique - this is an increase in the frequency of fragmentation with a lesion size of more than 20 mm, which in turn increases the risk of recurrence; with regard to ESD technique, this is a long procedure time; high incidence of complications; significant time required for teaching the technique; technical difficulties. In this regard, it is worth paying attention to the method of "endoscopic mucosal resection with circumferential mucosal incision" (C-EMR). This method deserves interest due to the fact that it allows more often to perform en-block resections in comparison with the classical method of endoscopic mucosal resection (EMR - endoscopic mucosal resection); technically easier to do; takes a short procedure time.

ELIGIBILITY:
Inclusion Criteria:

* patients with benign colon neoplasms without signs of deep invasion (I, II, IIIL and IV type according to Kudo, I and II type according to Sano)
* the size of the neoplasm is from 20 mm to 30 mm
* patient for treatment

Exclusion Criteria:

* unsatisfactory tumor lifting
* refusal of the patient from research at any stage of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-11-27 (Actual); Primary Completion 2023-09-27 (Estimated); Study Completion 2023-11-27 (Estimated)

PRIMARY OUTCOMES:
R0 resection rate | 14 day

SECONDARY OUTCOMES:
En-block resesction rate | 14 day
conversion rate | 1 day
intervention time | 1 day
intra- and postoperative complications rate | 30 day

CONTACTS AND LOCATIONS:
Locations (1):
- Elmira, Moscow, Russia